CLINICAL TRIAL: NCT05783687
Title: RWE Study of Subjects With Wilson's Disease to Assess Clinical Utility of Measuring Copper Parameters, Including a Novel Non-ceruloplasmin Bound Copper Assay Based on Copper Protein Speciation (NCC-Sp), Standard of Care Clinical and Biochemical Assessments
Brief Title: Real World Evidence Study in Subjects With Wilson's Disease
Acronym: REASON
Status: Completed | Type: Observational
Sponsor: Orphalan (Industry)
Responsible Party: Sponsor
Other Study IDs: ORPH-131-009
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-06

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Central laboratory blood samples taken for the study (i.e. not part of standard of care) may be kept for up to 5 years for additional testing (metal analyses). Up to 10mLs of blood should be collected for analysis of NCC-Sp, serum total copper and serum ceruloplasmin, copper fraction associated with ceruloplasmin and serum zinc levels at each study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- A - Newly diagnosed: Newly diagnosed (DPA/Trientine/Zinc for < 28 days)
  Interventions: Diagnostic Test: NCC-Sp Assay
- B - D-penicillamine: D-penicillamine
  Interventions: Diagnostic Test: NCC-Sp Assay
- C - Zinc: Zinc
  Interventions: Diagnostic Test: NCC-Sp Assay
- D - Trientine (2HCl or 4HCl): Trientine (2HCl or 4HCl)
  Interventions: Diagnostic Test: NCC-Sp Assay

INTERVENTIONS:
Diagnostic Test: NCC-Sp Assay — Orphalan has developed a new NCC speciation assay (NCC-Sp) using liquid chromatography inductively coupled plasma mass spectroscopy (LC-ICP-MS) to measure serum copper and ceruloplasmin bound copper from which non ceruloplasmin bound copper (NCC) is estimated.

SUMMARY:
This non-interventional Real-World Evidence (RWE) study aims to describe non-ceruloplasmin copper values obtained using a new NCC Speciation assay by taking a small (up to 10mLs) volume of additional blood from patients with Wilson's Disease, around the time when routine blood sampling is expected to be scheduled by the treating physician. Data will be collected over an approximate 12-month period.

DETAILED DESCRIPTION:
This is a non-interventional RWE study to describe NCC-Sp in relation to standard of care (SoC) copper measurements at each visit and longitudinally over an approximate 12-month study period in WD patients.

Data will be collected during routinely scheduled WD clinic visits over an approximate 12-month period.

Data collected will include:

* Relevant medical history and WD medication history
* All copper measurements and SoC clinical laboratory results prior to changing therapy/study enrolment, and if available, for up to 2 years prior to baseline
* Concomitant medications at the time of study enrollment and if available, for up to 2 years prior to baseline.
* Routine blood sample results from SoC assessments including biochemistry, hematology and coagulation measures, copper assessments (including serum ceruloplasmin and total copper alongside a locally calculated estimation of NCC).
* Around the same time as the routine blood samples, an additional study specific study blood samples of up to 10 mL will be collected for analysis of the NCC-Sp, serum total copper and serum ceruloplasmin, copper fraction associated with ceruloplasmin and serum zinc levels. Samples will be sent for analysis at the nominated central laboratory. Results will only be made available to investigators at the end of the study. Central laboratory samples taken for the study may be kept for up to 5 years for additional testing (metal analyses).
* Routine 24-hour urinary copper excretion (µmol/l) collection may form part of the SoC assessments conducted during regularly planned visits. This sample will be analyzed as per standard practice by the local laboratory.
* Calculated New Wilson's Disease Index and WD medications, and other testing as collected during routinely scheduled WD clinic visits and analyzed as per local hospital procedures and facilities.

After providing informed consent, patients meeting all inclusion and no exclusion criteria will be enrolled into the study. Patient's routine WD clinic visits will be scheduled according to the standard clinical practice at the study center and at the discretion of the treating physician. Enrolled patients are to be followed for approximately 12 months; first visit will be recorded as the baseline visit. If a switch of therapy is made, patients are typically re-assessed within a window of approximately 1- 3 months post initiation of the new treatment with biochemical testing and in person consultation for some. In the absence of starting a new treatment, patients are reviewed at approximately 6-month intervals, i.e., SoC visits at 6 months and 12 months. Routine chemistry, hematology, coagulation, copper assessments, 24h urine sampling for urinary copper excretion and other laboratory testing used to assess the patient as part of SoC will be performed as usual by the site local laboratory as determined by the treating physician per their standard practice for managing patients with WD. Routine safety testing and the required laboratory values produced by the local laboratory will be used to calculate the New Wilson's Disease Index.

An additional small volume (up to 10 mL) of blood will be drawn for central laboratory assessment of NCC-Sp, serum total copper and serum ceruloplasmin, copper fraction associated with ceruloplasmin and serum zinc levels around the same time as SoC blood draw is expected to minimize burden to the patients. These study specific samples will be drawn, processed, and shipped to a central laboratory either from the WD clinic, by a local commercial laboratory, or from the patient's home (or patient-specified local address) by a qualified home health care professional with experience in obtaining and processing blood specimens for clinical trials. Results from centrally processed samples will only be made available to investigators at the end of the study. Central laboratory samples taken for the study may be kept for up to 5 years for additional testing for metal analyses.

The following standardized disease assessment questionnaires will be conducted as per the schedule of assessments over the study:

* UWDRS (Part II)
* SF-12 quality of life questionnaire
* Morisky scale assessment for compliance (MMAS-8)
* Patient's Global Impression of Change (PGIC)
* Clinical Global Impression of Change (CGIC)

Central laboratory results (blood) will be transferred by the central laboratory vendor(s) for inclusion in the Clinical Data Set. The date of all sample collections as well as the results, units and normal range values from local laboratories and all other clinical data collected for the study (medical and medication history etc.) will be entered into a web-based electronic data capture (EDC) system by the study physician or study coordinator/designee.

Physicians are not obligated to actively seek information on adverse reactions/serious adverse reactions. However, if the Physician or other responsible person learns of any ADR /special reporting situation and he/she considers the event to be reasonably related to current treatment, the Investigator should document it in the eCRF. Adverse Drug Reactions attributable to a drug product, should be reported directly to the Marketing Authorisation Holder (MAH) of that product following the usual process.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent for participation in the study
2. Male or female patients, aged 18 years or older as of signing the Informed Consent Form (ICF)
3. Able and willing to comply with study procedures and requirements, as judged by the treating physician
4. Established diagnosis of Wilson's Disease (Leipzig score >4)
5. Either newly diagnosed or with elevated liver enzymes (defined as ALT, AST ≥1.5xULN) or 24-hour urinary copper excretion outside of recommended ranges [chelation range 200-500mcg/24 hr; zinc < 100mcg/24 hr]
6. Adequate venous access to allow collection of blood samples

Exclusion Criteria:

1. Major systemic disease or other illness that would, in the opinion of the investigator, compromise patient safety or interfere with the collection or interpretation of the study results.
2. Patients with a New Wilson's Disease Index Score of >7
3. In the opinion of the investigator, the patient is likely to be non-compliant or uncooperative for routine clinical visits during the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 18 years old) with Wilson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
The distribution of Non-Ceruloplasmin bound Copper (NCC) in serum as assessed by a NCC-speciation LC-ICP-MS assay (NCC-Sp), at study entry and over an approximate 12-month period from a real-world population of WD patients. | Approx 12 Months
  The distribution of NCC-Sp will be assessed as a diagnostic value, to be used for adjusting chelation therapy in Wilson Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Schilsky, Principal Investigator — Yale University School of Medicine, New Haven, Connecticut
Locations (9):
- United States (9):
  - UC Davis Midtown Ambulatory Care Centre, Sacramento, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Northwestern University Chicago (Hepatologist), Chicago, Illinois
  - John Hopkins Hospital, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - New York Presbyterian Hospital-Columbia University Medical Centre, New York, New York
  - Vanderbilt University Medical Centre, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided